CLINICAL TRIAL: NCT05666960
Title: A Single and Repeat Dosing Study of the Safety, Drug Exposure, and Clinical Activity of R-3750 in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: R-3750 in Patients With Mild to Moderate Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rise Therapeutics LLC (Industry)
Collaborators: Mayo Clinic (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISE R-3750-01
Record Dates: First submitted 2022-12-01; First posted 2022-12-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate; Ulcerative Colitis Chronic; Ulcerative Colitis
Keywords: Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: R-3750 — Probiotic

SUMMARY:
The goal of this study is to determine the safety and tolerability of orally taken probiotic (R-3750) in patients with mild to moderate ulcerative colitis.

Patients will take an oral dosage of probiotic (R-3750) and provide patient-reported and physician scored measures of their colitis. Blood and fecal evaluations of inflammation and assessment of probiotic (R-3750) on fecal levels will also be measured.

ELIGIBILITY:
INCLUSION CRITERIA:

* 18-65 years of age
* Ability to provide written informed consent
* Confirmed diagnosed with UC by colonoscopy and histology and suffering from mild to moderate UC as defined by MMDAI with score of 3-9
* On a stable dose of aminosalicylate (i.e. no change in medication within 4 weeks of study enrollment) and not planning to initiate new medication other than the study drug
* For women of childbearing potential or men with a partner of childbearing potential, agree to use birth control methods (including hormonal contraceptives, intrauterine device (IUD) or hormone releasing system (IUS), vasectomy) and men will refrain from donating sperm during the study and at least 30 days after dosing (per FDA guidelines)
* For the expansion cohort, a flexible sigmoidoscopy is required, unless an endoscopy was completed within 3 months from enrollment is available
* Refrain from receiving any type of vaccinations during the study period (to include but not limited to influenza, COVID, shingles, tetanus, hepatitis, pneumonia, HPV, DPT, MMR, and polio)

EXCLUSION CRITERIA:

* Pregnancy, planned pregnancy, breastfeeding women
* Evidence of severe UC disease (MMDAI score greater than or equal to 10)
* Evidence of any active or recent infection including chronic infectious disease such as Hepatitis B, C, or HIV
* Evidence of any active or recent chronic chest infection with bronchiectasis or sinusitis, or covid-19 infection in the past 3 months
* Treatment with immunosuppressants or anti-cancer drugs, e.g., anti-TNF-α agents, anti-integrin agents, azathioprine or 6-MP, 6-thioguanine, methotrexate, ozanimod, tofacitinid, upadacitinib, tacrolimus, cyclophosphamide, or cyclosporine or any other therapy that is not an aminosalicylate within the last 3 months
* Received an investigational drug within 3 months (or 5 half-lives, whichever is longer) before study entry
* Use of steroidal drugs to treat UC (e.g., prednisone >20 mg/day)
* Use of probiotics within the last one (1) week and during the trial.
* Treatment with systemic broad-spectrum antibiotics in the past 2 months
* Major active systemic autoimmune disease other than UC
* History of anaphylaxis or allergies to probiotics
* History of alcohol or drug abuse within the past 2 years
* History of stroke, or any cerebrovascular disease requiring medication/treatment
* History of cancer, apart from successfully treated basal cell carcinoma or in situ carcinoma of the cervix >1 year prior to enrollment
* Significant laboratory abnormalities, including liver transaminases (AST or ALT) > 1.5X the upper limit of normal.
* Second degree or higher heart block or clinically significant arrythmia
* Any other clinically significant renal, hepatic, hematological or other disease or laboratory abnormality which, in the opinion of the investigator, would interfere with the conduct, the interpretation of the safety signals or results of the trial, or would place the subject at unacceptable risk
* Any condition or circumstance that, in the opinion of the Principal Investigator, would compromise the safety of the subject or the quality of study data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess the tolerability of R-3750 | 6 weeks
  To assess the number of participants with treatment-realated adverse events after taking R-3750 (probiotic)

SECONDARY OUTCOMES:
Clinical Response based on Inflammatory Bowel Disease Questionnaire (IBDQ) Scores | 6 weeks
  To assess the number of participants that show improvements in the ulcerative colitis disease severity by collecting IBDQ. The scores are based on a numbering system from one (1) to seven (7) where seven (7) is the least about of trouble with your bowels and one (1) is the most. The numbers are totaled to provide a total score from 32 to 224. Where 32 is a better outcome and 224 is a worse outcome. This is compared from the beginning and again at different times to see if there are any changes to your microbiome before and after taking R-3750 (probiotic).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Amicis Research Center, Valencia, California
  - AP Medical Research LLC, Miami, Florida
  - Edward Jenner Research Group, LLC, Plantation, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided